CLINICAL TRIAL: NCT03523364
Title: Long -Term Survival Rate of All Ceramic Restorations Cemented With Air-Water-Blasting Treatment Compared to Control Treatment
Brief Title: Survival Rate of All Ceramic Restorations Treated With Air-Water-Blasting Protocol
Status: Completed | Type: Observational
Sponsor: Università degli Studi 'G. d'Annunzio' Chieti e Pescara (Other)
Responsible Party: Principal Investigator, Traini Tonino, senior researcher, Università degli Studi 'G. d'Annunzio' Chieti e Pescara
Other Study IDs: 84183
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Survival, Prosthesis
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: dental restorations — partial or complete ceramic restorations bonded to dental tissues after WAB and total etching or after total etching

SUMMARY:
This study evaluates retrospectively the survival rate of all-ceramic restorations, cemented using AWB technique (test) compared to those cemented with conventional technique (control)

DETAILED DESCRIPTION:
A retrospective study on ceramic restorations, placed in the period 2003-2014, will be performed to assess the survival rate of all-ceramic restorations cemented adhesively. The effectiveness of cementation largely depend on the method used. The Air-Water-blasting performed prior to conventional acid-etch of dental tissues offers an increase in bond strength compared to the conventional etching technique.

ELIGIBILITY:
Inclusion Criteria:

* patients who received at least one ceramic restoration

Exclusion Criteria:

* patients who received feldspathic ceramic restorations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients treated for bonded all-ceramic restorations between years 2003-2014
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
survival rate | 2003-2014
  integrity of the restorations

CONTACTS AND LOCATIONS:
Overall Officials: Tonino Traini, DDS; PhD, Principal Investigator — University of Chieti-Pescara
Locations (1):
- Dipartimento di Scienze Mediche Orali e Biotecnologiche, Chieti, CH, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van den Breemer CR, Vinkenborg C, van Pelt H, Edelhoff D, Cune MS. The Clinical Performance of Monolithic Lithium Disilicate Posterior Restorations After 5, 10, and 15 Years: A Retrospective Case Series. Int J Prosthodont. 2017 Jan/Feb;30(1):62-65. doi: 10.11607/ijp.4997. PMID 28085983
- [Background] Beier US, Kapferer I, Dumfahrt H. Clinical long-term evaluation and failure characteristics of 1,335 all-ceramic restorations. Int J Prosthodont. 2012 Jan-Feb;25(1):70-8. PMID 22259801